CLINICAL TRIAL: NCT02938936
Title: Waiting Time. Wasting Time: A Randomized Control Trial to Investigate the Health Impacts of Improving the Quality of Antenatal Care in Mozambique
Brief Title: Waiting Time. Wasting Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: London School of Economics and Political Science (Other)
Responsible Party: Principal Investigator, Margaret McConnell, Assistant Professor of Global Health Economics, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0344
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scheduling Intervention (Experimental): Pre-natal visit scheduling
  Interventions: Other: Pre-natal visit scheduling
- Control (No Intervention)

INTERVENTIONS:
Other: Pre-natal visit scheduling — This intervention will include a scheduled date and time for prenatal care follow-up visits. Women in the intervention group seeking care for their first ANC appointment will be offered several appointment slots on their return date by the nurse providing their first ANC visit. Women will be able select among the time options and will be provided an appointment card with their scheduled date and time. Staff will limit the number of scheduled women per hour by maintaining an appointment book. Clinic staff will be trained to differentiate between women returning for a scheduled visit from first prenatal visits, emergencies, and unscheduled return visits. First visits and emergencies will be seen during the first 2 hours after clinic opening and unscheduled women will be seen during a one-hour time slot midday. When women return on their date, they will be seen within one hour of their appointment time by clinic staff.
  Arms: Scheduling Intervention

SUMMARY:
Our study's principle purpose is to determine whether decreasing waiting time before being seen for antenatal care increases demand for and use of antenatal care services in Mozambique.

DETAILED DESCRIPTION:
This protocol describes a pilot study that will test the impact of a scheduling intervention intended to reduce waiting times for antenatal care. The study will include one intervention health clinic and one control clinic in Maputo, Mozambique. In the intervention facility women attending antenatal care will be informed that if they return at their scheduled date and time they will be seen within one hour by clinic staff rather than having to wait for an indefinite amount of time before being seen for care. Appointment cards will be clipped into ANC cards, which collect routine health data and are kept by women at the end of their ANC visit. Health facility staff will be trained to identify women who return at their scheduled time and to manage patient flow such that scheduled women are received quickly. After the start date of the intervention, all women attending ANC at the health facility will be provided a scheduled return date and time window. Baseline and endline exit interview surveys will be conducted in both intervention and control facilities to compare changes in waiting time, number of ANC visits, and provider satisfaction over the course the study period between clinics.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for individual study participants enrolled after delivery:

1. Women who delivered at the health facility during the weeks of recruitment

Inclusion criteria for women whose waiting time is measured:

1. Women at the health facility to seek care for antenatal care or another reproductive health service (anticipate total enrollment of 800 women)

Inclusion criteria for the health care provider survey is that the provider

1. Have worked in the health facility for at least 6 months
2. The health care worker provides ANC as part of their routine duties (anticipate total enrollment of 4 health care workers)

Exclusion Criteria:

Exclusion criteria for individual study participants enrolled after delivery:

1. Women under 18 years of age will be excluded
2. Women whose babies die during labor or childbirth from the delivery exit interviews

There are no exclusion criteria for the sample of women whose waiting time will be measured There are no exclusion criteria for the health care provider survey

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in percent of women completing at least 4 prenatal care visits before and after intervention | During most recent pregnancy, as reported in an exit survey conducted at discharge from delivery at baseline and six months after the start of the scheduling intervention
Change in average waiting time before being seen for prenatal care before and after intervention | Measured for 4 weeks at baseline before the start of the intervention, and for 4 weeks, 3 months after the start of the intervention

SECONDARY OUTCOMES:
Change in nurses satisfaction with their job (1-5 scale) | Measured before the start of the intervention, and 6 months after the start of the intervention
Change in proportion of key ANC services respondent reports receiving at most recent prenatal care visit, 9 possible services measured in exit survey at discharge from delivery. | Measured at baseline and 6 months after the start of the intervention
  9 key services include:
  * IPTP dose provided, measured by self-report
  * Delivery plan discussed, measured by self-report
  * Hemoglobin test measured by patient report of having had their blood drawn
  * Recommendations for family planning and breast feeding provided, measured by self-report
  * Detection of breech measured by report of the provider palpating the tummy
  * Blood pressure
  * Measurement of uterine height
  * Urine test
  * Recommendation for what to do in emergencies

REFERENCES:
- [Derived] Steenland M, Dula J, de Albuquerque A, Fernandes Q, Cuco RM, Chicumbe S, Gudo ES, Sequeira S, McConnell M. Effects of appointment scheduling on waiting time and utilisation of antenatal care in Mozambique. BMJ Glob Health. 2019 Nov 25;4(6):e001788. doi: 10.1136/bmjgh-2019-001788. eCollection 2019. PMID 31803509